CLINICAL TRIAL: NCT02209662
Title: A Multi-Center, Randomized Trial Comparing the Effectiveness of APIC-PRP to Control, When Added to Standard of Care in the Treatment of Non-healing Diabetic Foot Ulcers
Brief Title: Safety and Efficacy Study of APIC-PRP in Non-healing Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cytonics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cyt201-01
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Diabetic Foot Ulcer
Keywords: APIC-PRP; Chronic Wounds; Diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Sodium Chloride; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- APIC-PRP and Standard of Care (Experimental): APIC-PRP
  Interventions: Device: APIC-PRP
- Placebo, Saline plus standard of care (Placebo Comparator): Placebo, Saline plus standard of care
  Interventions: Other: Placebo, Saline plus standard of care

INTERVENTIONS:
Device: APIC-PRP — APIC-PRP
  Arms: APIC-PRP and Standard of Care
Other: Placebo, Saline plus standard of care — Placebo, Saline plus standard of care
  Arms: Placebo, Saline plus standard of care

SUMMARY:
Patients have a diabetic foot ulcer that is older than 4 weeks and has been treated with physician-selected standard of care treatment such as debridement, hydrogel or saline irrigation, primary dressing, and offloading will be randomized into one of two groups, the Standard of Care (SoC) or APIC-PRP + SoC. APIC-PRP has high level of platelets that produce growth factors that can help in wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Prior to the first clinical intervention, a signed Informed Consent Form (ICF) and Data Consent Form (DCF) must be obtained from the subject or legal representative
* Diagnosed with insulin-dependent or non-insulin-dependent diabetes (Type I or II, respectively), requiring medical treatment as determined by the physician
* Subjects will have only one diabetic foot ulcer on the target limb (referred to as the Index Ulcer)
* The Index Ulcer, classified using the University of Texas Wound Classification System (Appendix 7), is located on the dorsal, plantar, medial, or lateral aspect of the foot or heel (including all toe surfaces)
* Debrided ulcer size between 1 cm2 and 4 cm2. See Appendix 3 for instructions on wound area measurement
* DFU with a duration ≥ 1 month at first visit
* The target ulcer is free of clinical signs of infection, identified by inflammation (redness, warmth, swelling, tenderness, or pain) or purulent exudates (Lipsky et al, 2012).
* The patient meets Medicare/Medicaid eligibility requirements. Subject's ulcer extends through the dermis and into subcutaneous tissue (granulation tissue may be present) but without exposure of muscle, tendon, bone or joint capsule.
* Post-debridement, subject's wound is free of necrotic debris and appears to be made up of healthy vascularized tissue.
* Demonstrated adequate offloading regimen.
* Subject has adequate circulation to the study foot as evidenced by a Doppler measured ankle-bronchial index (ABI) of ≥ 0.7 after 10 minutes of rest
* Age >18 years old at the time the informed consent is signed
* Female subjects must have a negative urine pregnancy test prior to the first treatment
* Subject must be willing to comply with the Protocol, which will be assessed by enrolling clinician

Exclusion Criteria:

* Subject has inadequate venous access the blood draw required for APIC-PRP Administration. Subjects with PIC or IV access are preferred.
* Hemoglobin of less than 12 g/dL
* Inadequate amount of blood drawn to produce sufficient APIC-PRP. One complete APIC-PRP preparation requires 114ml of blood drawn per APIC-PRP preparation.
* Subject's ulcer has increased in size by >50% during the run-in Screening period.
* If the subject's ulcer healed by 25% or more during the run-in Screening period they will be excluded.
* Presence of another wound that is concurrently treated and might interfere with treatment of the index wound by APIC-PRP (malignancy in nearby wound)
* Ulcer not of DFU pathophysiology (e.g., venous, vasculitic, radiation, rheumatoid, collagen vascular disease, pressure, or arterial etiology)
* The target ulcer demonstrates underlying osteomyelitis, defined as infection in the bone, identified by Fever, chills, or pain in the infected bone. Any exposed bone will be classified as osteomyelitis.
* Subject has a history of bleeding disorder.
* Any malignancy other than non-melanoma skin cancer requiring treatment with immunosuppressive or chemotherapeutic agents, radiotherapy or corticosteroids less than 30 days before enrolment.
* Subject has gangrene present on any part of the affected limb. Subject's ulcer is over a Charcot deformity of the mid-foot ("Rocker-Bottom Foot") or over the tarsal bones-talus, distal calcaneus, navicular, and cuboid.
* Subject's ulcer has tunnels or sinus tracts that cannot be completely debrided.
* Subject has severe malnutrition as evidenced by albumin < 2.5 g/dL. A previous serum albumin test that is <6 weeks old is sufficient for this criteria.
* Subject has Acquired Immunodeficiency Syndrome (AIDS), liver disease, aplastic anemia, scleroderma, malignancy, cellulitis, suspected osteomyelitis or other evidence of systemic infection, or is Human Immunodeficiency Virus (HIV)-positive.
* Subject has any elective osseous procedures to the study foot within 30 days prior to the Initial Visit.
* Subject is on dialysis.
* Subjects who are cognitively impaired and therefore can not give consent, and do not have a healthcare proxy
* Subjects who, in the opinion of the Investigator, represent poor medical, psychological or psychiatric risks for whom therapy with an investigational product would be unwise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Complete wound closure within 12 weeks | 12 weeks
  The primary outcome expected for this study is an increase in the proportion of DFUs that have exhibited complete closure within 12 weeks between the APIC-PRP + SoC groups and SoC alone groups.

SECONDARY OUTCOMES:
Improvement in wound healing trajectory within 12 weeks | 12 weeks
  The secondary outcome expected for this study is an improvement in wound healing trajectory of DFUs over the 12 weeks treatment period between the APIC-PRP + SoC groups and SoC alone groups.
Improvement in wound healing for the patient to return to function over the 12 weeks | 12 weeks
  The secondary outcome expected for this study is an improvement in wound healing for the patient to return to function over the 12 weeks treatment period between the APIC-PRP + SoC groups and SoC alone groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano J Scuderi, MD, Study Director — Cytonics Corporation